CLINICAL TRIAL: NCT05531565
Title: A 2-Part Seamless Part A (Phase 2)/Part B (Phase 3) Randomized, Double-Blind, Placebo-Controlled, Multicenter Study to Evaluate the Efficacy and Safety of BIIB059 in Participants With Active Subacute Cutaneous Lupus Erythematosus and/or Chronic Cutaneous Lupus Erythematosus With or Without Systemic Manifestations and Refractory and/or Intolerant to Antimalarial Therapy (AMETHYST)
Brief Title: A 2-Part Study to Learn Whether Litifilimab (BIIB059) Injections Can Improve Symptoms of Adult Participants Who Have Active Cutaneous Lupus Erythematosus
Acronym: AMETHYST
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 230LE301; 2020-000727-40 (EudraCT Number); EU CT Number (Other: 2023-505634-94-00)
Record Dates: First submitted 2022-08-19; First posted 2022-09-08 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Subacute Cutaneous Lupus Erythematosus; Chronic Cutaneous Lupus Erythematosus
Keywords: Cutaneous Lupus Erythematosus (CLE); Acute Cutaneous Lupus Erythematosus (ACLE); Discoid Lupus Erythematosus (DLE); Systemic Lupus Erythematosus (SLE); Lupus
MeSH Terms: conditions — Lupus Erythematosus, Cutaneous; Lupus Erythematosus, Discoid; Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Part A (Phase 2): Litifilimab (Experimental): Participants will receive litifilimab subcutaneously (SC) once every 4 weeks (Q4W) from Week 0 to Week 20, with an additional dose of litifilimab at Week 2 during the double-blind placebo-controlled (DBPC) treatment period. Following the DBPC treatment period, participants will receive litifilimab during the extended treatment period (ETP) from Week 24 to Week 48, with an additional dose of litifilimab-matching placebo at Week 26.
  Interventions: Drug: Litifilimab
- Part A (Phase 2): Placebo (Placebo Comparator): Participants will receive litifilimab-matching placebo SC Q4W from Week 0 to Week 20, with an additional dose of litifilimab-matching placebo at Week 2 during the DBPC treatment period. Following the DBPC treatment period, participants will receive litifilimab during the ETP from Week 24 to Week 48, with an additional dose of litifilimab at Week 26.
  Interventions: Drug: Placebo
- Part B (Phase 3): Litifilimab (Experimental): Participants will receive litifilimab SC Q4W from Week 0 to Week 20, with an additional dose of litifilimab at Week 2 during the DBPC treatment period. Following the DBPC treatment period, participants will receive litifilimab during the ETP from Week 24 to Week 48, with an additional dose of litifilimab-matching placebo at Week 26.
  Interventions: Drug: Litifilimab
- Part B (Phase 3): Placebo (Placebo Comparator): Participants will receive litifilimab-matching placebo SC Q4W from Week 0 to Week 20, with an additional dose of litifilimab-matching placebo at Week 2 during the DBPC treatment period. Following the DBPC treatment period, participants will receive litifilimab during the ETP from Week 24 to Week 48, with an additional dose of litifilimab at Week 26.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Litifilimab — Administered as specified in the treatment arm.
  Other Names: BIIB059
  Arms: Part A (Phase 2): Litifilimab; Part B (Phase 3): Litifilimab
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Part A (Phase 2): Placebo; Part B (Phase 3): Placebo

SUMMARY:
In this study, researchers will learn more about a study drug called litifilimab (BIIB059) in participants with cutaneous lupus erythematosus (CLE). The study will focus on participants who have either active subacute CLE or chronic CLE, or both. They may also have systemic lupus erythematosus (SLE). The participants did not respond to antimalarial therapy or had problems with the treatment that made it hard to continue.

The main objective of the study is to learn about the effect litifilimab has on lowering the activity of the skin disease. Researchers will measure symptoms of CLE over time using a variety of scoring tools. These include the Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI), the Cutaneous Lupus Activity of Investigator's Global Assessment-Revised (CLA-IGA-R), and the SELENA-SLEDAI Flare Index (SFI).

The main questions researchers want to answer are:

* How many participants have a score of 0 or 1 on the CLA-IGA-R looking at skin redness after treatment?
* How many participants have their skin disease activity go down by at least 70%?

Researchers will also learn more about the safety of litifilimab. They will study how participants' immune systems respond to litifilimab. Additionally, they will measure the effect litifilimab and CLE have on the quality of life of participants using a group of questionnaires.

The study will be split into 2 parts - Part A and Part B. Both parts will be done as follows:

* After screening, participants will be randomized to receive either litifilimab or placebo for the 1st treatment period. A placebo looks like the study drug but contains no real medicine.
* Participants will receive either litifilimab or placebo as injections under the skin once every 4 weeks.
* The 1st treatment period will be double blinded which means neither the researchers nor the participants will know if the participants are receiving litifilimab or placebo.
* This double blinded treatment period will last 24 weeks, after which the 2nd treatment period will begin.
* During the 2nd treatment period, all participants will receive litifilimab for 28 weeks.
* After completing treatment in this study, participants that qualify will be given the choice to join the Long-Term Extension study, 230LE305. If they do not, they will move into a follow-up safety period that will last up to 24 weeks.
* The total study duration for participants will be up to 80 weeks

DETAILED DESCRIPTION:
Litifilimab is a humanized immunoglobulin G1 (IgG1) monoclonal antibody targeting blood dendritic cell antigen 2 and is being investigated for the potential treatment of systemic lupus erythematosus and cutaneous lupus erythematosus. The primary objectives of the study are to evaluate the efficacy of litifilimab compared with placebo in reducing skin disease activity measured by the CLA-IGA-R score [Parts A and B (US)] and the Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity (CLASI-A) score [Part B (ROW)] in participants with active SCLE and/or CCLE with or without systemic manifestations and refractory and/or intolerant to antimalarials. The secondary objectives of the study are to evaluate the efficacy of litifilimab in reducing SCLE and/or CCLE disease activity by CLA-IGA-R, CLASI-A; to evaluate additional efficacy parameters of litifilimab in reducing SCLE and/or CCLE disease activity; safety; tolerability; and immunogenicity of litifilimab [Parts A and B].

ELIGIBILITY:
Key Inclusion Criteria:

1. Histologically confirmed (in the past or during the Screening period) diagnosis of CLE with or without systemic manifestations.
2. Must have active cutaneous manifestations that meet study criteria.
3. Must have a CLASI-A score ≥10.
4. Must have an active CLE lesion despite an adequate trial of antimalarial treatment.

Key Exclusion Criteria:

1. Any active skin conditions other than CLE that may interfere with the study assessments of CLE.
2. Diagnosis of mixed connective tissue disease [(within 1 year of signing the informed consent form (ICF)] or any history of overlap syndromes of SLE including concomitant presence with rheumatoid arthritis, dermatomyositis and/or polymyositis, systemic sclerosis, psoriatic arthritis, or any other autoimmune disease that may confound the evaluation of the disease activity or the effect of the investigational product. Exceptions for overlap syndrome of SLE include participants with overlap syndrome of SLE with myositis and secondary Sjögren's syndrome at screening is permitted provided the participant also meets the criteria for classification as SLE. A past history of mixed connective tissue disease that over time has developed into a diagnosis of SLE is permitted, provided diagnosis of SLE has been present for at least 1 year.
3. Active severe lupus nephritis.
4. Active neuropsychiatric SLE.
5. Use of intralesional corticosteroids within 1 week prior to Screening and during the study.
6. Use of immunosuppressive or disease-modifying treatments for SLE or CLE [via an oral, intravenous (IV), or SC route] that were initiated less than 12 weeks prior to randomization, have not been at a stable and allowable dose.

NOTE: Other protocol-defined Inclusion/Exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 474 (Estimated)
Dates: Start 2022-09-13 (Actual); Primary Completion 2026-10-20 (Estimated); Study Completion 2027-12-14 (Estimated)

PRIMARY OUTCOMES:
Parts A (US+ROW) and B (US): Percentage of Participants who Achieve a Cutaneous Lupus Activity of Physician's Global Assessment-Revised (CLA-IGA-R) Erythema Score of 0 or 1 | Week 16
Part B (ROW): Percentage of Participants who Achieve Cutaneous Lupus Erythematosus Disease Area and Severity Index Activity Score (CLASI-70) Response, Defined as ≥ 70% Decrease in CLASI-A Score From Baseline | Baseline to Week 24

SECONDARY OUTCOMES:
Part A (US+ROW): Percentage of Participants who Achieve a CLASI-50 Response, Defined as a ≥ 50% Decrease in CLASI-A Score From Baseline | Weeks 16 and 24
Part A (US+ROW): Absolute Change in Cutaneous Lupus Erythematosus Disease Area and Severity Index Damage (CLASI-D) Score at Week 52 | Baseline to Week 52
Part A (US+ROW): Percent Change in CLASI-D Score | Baseline to Week 52
Part B (US+ROW): Percentage of Participants who Achieve a CLA-IGA-R Erythema Score of 0 or 1, at Week 16 and Week 24, Respectively, for Participants in Full Analysis Set (FAS), who had CLA-IGA-R Erythema Score ≥3 and Other OMC Score ≥3 at Baseline | Weeks 16 and 24
Part B (US+ROW): Percentage of Participants who Achieve a CLA-IGA-R OMC Score of 0 or 1, at Week 16 and Week 24, Respectively, for Participants in FAS, who had CLA-IGA-R Erythema Score ≥3 and OMC Score ≥3 at Baseline | Weeks 16 and 24
Part B (US+ROW): Percentage of Participants who Achieve at Least 1 Level of Improvement From Baseline in the CLA-IGA-R Erythema Score | Up to Week 24
Part B (US+ROW): Absolute Change in CLASI-D Score | Week 52
Part B (US+ROW): Percent Change in CLASI-D Score | Week 52
Part B (US+ROW): Change From Baseline in Cutaneous Lupus Erythematosus-Quality of Life (CLE-QoL) Score | Part B (US): Weeks 16 and 52; Part B (ROW): Weeks 24 and 52
Part B (US+ROW): Change From Baseline in Dermatology Life Quality Index (DLQI) Score | Part B (US): Weeks 16 and 52; Part B (ROW): Weeks 24 and 52
Part B (US+ROW): Change From Baseline in Numerical Rating Scale (NRS) for Pain in Skin Rash | Part B (US): Weeks 16 and 52; Part B (ROW): Weeks 24 and 52
Part B (US+ROW): Change From Baseline in NRS for Itch in Skin Rash | Part B (US): Weeks 16 and 52; Part B (ROW): Weeks 24 and 52
Parts A (US+ROW) and B (US): Percentage of Participants who Achieve a CLASI-70 Response, Defined as a ≥ 70% Decrease in CLASI-A Score From Baseline | Part A (US+ROW): Weeks 16 and 24; Part B (US): Week 16
Parts A and B (US+ROW): Percentage of Participants who Achieve a CLA-IGA-R Erythema Score of 0 or 1 | Part A (US+ROW): Week 24; Part B (ROW): Week 24; Part B (US+ROW): Up to Week 24
Parts A and B (US+ROW): Percentage of Participants who Achieve a CLA-IGA-R Other Morphologic Characteristics (OMC) Score of 0 or 1 and at Least 1 Level of Improvement From Baseline | Part A (US+ROW): Weeks 16 and 24; Part B (US): Week 16; Part B (ROW): Week 24; Part B (US+ROW): Up to Week 24
Parts A and B (US+ROW): Percentage of Participants who Achieve a CLA-IGA-R OMC Score of 0 | Part A (US+ROW): Weeks 16 and 24; Part B (US+ROW): Up to Week 24
Parts A and B (US+ROW): Percentage of Participants With at Least 1 Level of Improvement From Baseline in CLA-IGA-R OMC Score | Part A (US+ROW): Weeks 16 and 24; Part B (US+ROW): Up to Week 24
Parts A and B (US+ROW): Percentage of Participants who Achieve a CLA-IGA-R Follicular Activity Score of 0 | Parts A and B (US+ROW): Weeks 16 and 24; Part B (US+ROW): Up to Week 24
Parts A and B (US+ROW): Percentage of Participants who Achieve a CLASI-A Score of 0 or 1 | Up to Week 24
Parts A and B (US+ROW): Percentage of Participants who Achieve a CLASI-A Score of 0 to 3 | Up to Week 24
Parts A and B (US+ROW): Percentage of Participants who Achieve a CLASI 70 Response | Up to Week 24
Parts A and B (US+ROW): Percentage of Participants who Achieve a CLASI 50 Response | Up to Week 24
Parts A and B (US+ROW): Percentage of Participants who Achieve a 7-Point Reduction From Baseline in CLASI-A Score | Up to Week 24
Parts A and B (US+ROW): Percentage of Participants With a CLASI-70 Response at Week 52 Among CLASI-70 Responders at Week 16 and Week 24, Respectively, who Were Randomly Assigned to Receive Litifilimab During the DBPC Treatment Period (TP) | Week 52
Parts A and B (US+ROW): Percentage of Participants With CLA-IGA-R Erythema Score of 0 or 1 at Week 52 Among CLA-IGA-R Erythema Responders at Week 16 and Week 24, Respectively, who Were Randomly Assigned to Receive Litifilimab During the DBPC TP | Week 52
Parts A and B(US+ROW): Percentage of Participants With CLA-IGA-R OMC Score of 0/1 & at Least 1 Level of Improvement From Baseline at Week 52 Among CLA-IGA-R OMC Responders at Weeks 16 &24, Respectively, who Were Assigned to Receive Litifilimab in DBPC TP | Week 52
Parts A and B (US+ROW): Percentage of Participants With CLA-IGA-R OMC Score of 0 at Week 52 Among CLA-IGA-R OMC Responders With CLA-IGA-R OMC Score of 0 at Week 16 and Week 24, Respectively, who Were Randomly Assigned to Litifilimab During DBPC TP | Week 52
Parts A and B(US+ROW):Percentage of Participants With CLA-IGA-R Follicular Activity Score of 0 at Week 52 Among CLA-IGA-R Follicular Activity Responders at Week 16 and Week 24, Respectively, who Were Randomly Assigned to Receive Litifilimab in DBPC TP | Week 52
Parts A and B (US+ROW): Percentage of Participants With a CLASI-70 Response at Week 52 Among CLASI-70 Nonresponders at Week 16 and Week 24, Respectively, who Were Randomly Assigned to Receive Placebo During the DBPC TP | Week 52
Parts A and B (US+ROW): Percentage of Participants With a CLA-IGA-R Erythema Score of 0 or 1 at Week 52 Among CLA-IGA-R Erythema Nonresponders at Week 16 and Week 24, Respectively, who Were Randomly Assigned to Receive Placebo During the DBPC TP | Week 52
Parts A, B(US+ROW):Percentage of Participants With CLA-IGA-R OMC Score of 0/1 and at Least 1 Level of Improvement From Baseline at Week 52 Among CLA-IGA-R OMC Nonresponders at Weeks 16 and 24, Respectively, who Were Assigned to Receive Placebo in DBPC TP | Week 52
Parts A and B (US+ROW): Number of Participants With Anti-Litifilimab Antibodies in Serum During the Study | Up to Week 76
Parts A and B (US+ROW): Percentage of Participants With a CLA-IGA-R OMC Score of 0 at Week 52 Among CLA-IGA-R OMC Nonresponders at Week 16 and Week 24, Respectively, who Were Randomly Assigned to Receive Placebo During the DBPC TP | Week 52
Parts A and B(US+ROW): Percentage of Participants who Achieve CLA-IGA-R Follicular Activity Score of 0 at Week 52 Among CLA-IGA-R Follicular Activity Nonresponders at Weeks 16 and 24, Respectively, who Were Randomly Assigned to Receive Placebo in DBPC TP | Week 52
Parts A and B (US+ROW): Annualized Mild and Moderate Safety of Estrogens in Lupus Erythematosus National Assessment-SLE Disease Activity Index Flare Index (SFI) Rate and Annualized Severe SFI Rate Through Week 24 | Up to Week 24
Parts A and B (US+ROW): Annualized Mild and Moderate SFI Rate and Annualized Severe SFI Rate Through Week 16 | Up to Week 16
Parts A and B (US+ROW): Annualized Mild and Moderate SFI Rate and Annualized Severe SFI Rate Through Week 52 | Up to Week 52
Parts A and B (US+ROW): Number of Participants Experiencing Treatment Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to Week 76

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (289):
- United States (61):
  - Pinnacle Research Group, LLC, Anniston, Alabama
  - UAB Center for Women's Reproductive Health, Birmingham, Alabama
  - Arizona Arthritis & Rheumatology Research, PLLC, Phoenix, Arizona
  - The Regents of the University of California, La Jolla, California
  - Dermatology Research Associates, Los Angeles, California
  - Clinical Science Institute, Santa Monica, California
  - Inland Rheumatology Clinical Trials, Inc., Upland, California
  - Denver Arthritis Clinic, Denver, Colorado
  - Omega Research Debary, LLC, DeBary, Florida
  - Centre for Rheumatology, Immunology and Arthritis, Fort Lauderdale, Florida
  - University of Florida, Gainesville, Florida
  - University of Miami Miller School of Medicine, Miami, Florida
  - Millennium Medical Research, LLC, Miami, Florida
  - Medical Research Center of Miami, Miami, Florida
  - Diverse Clinical Research LLC, Miami, Florida
  - Charisma Medical and Research Center, Miami Lakes, Florida
  - Leading Edge Dermatology, Plantation, Florida
  - Augusta University, Augusta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - OrthoIllinois, Rockford, Illinois
  - Dawes Fretzin Clinical Research Group, LLC, Indianapolis, Indiana
  - Equity Medical, Bowling Green, Kentucky
  - LSU Health Sciences Center Shreveport, New Orleans, Louisiana
  - Tufts Medical Center, Boston, Massachusetts
  - Brigham And Women's Hospital, Boston, Massachusetts
  - Essential Dermatology, Natick, Massachusetts
  - Beacon Clinical Research, LLC, Quincy, Massachusetts
  - University of Massachusetts, Worcester, Worcester, Massachusetts
  - David Fivenson, MD, Dermatology, PLLC, Ann Arbor, Michigan
  - Oakland Hills Dermatology, Auburn Hills, Michigan
  - AA MRC LLC Ahmed Arif Medical Research Center, Flint, Michigan
  - Revival Research Institute, LLC, Troy, Michigan
  - Saint Louis University, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Albuquerque Center For Rheumatology, Albuquerque, New Mexico
  - University of New Mexico School of Medicine, Albuquerque, New Mexico
  - NYU Langone Brooklyn, Brooklyn, New York
  - Universal Dermatology, PLLC, Fairport, New York
  - Northwell Health, Inc. PRIME, Great Neck, New York
  - Columbia University Medical center, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke Dermatology South Durham, Durham, North Carolina
  - Medication Management, LLC, Greensboro, North Carolina
  - University of Cincinnati Department of Dermatology, Cincinnati, Ohio
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - Penn State University Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Austin Regional Clinic, P.A., Austin, Texas
  - Precision Comprehensive Clinical Research Solutions, Colleyville, Texas
  - Metroplex Clinical Research Center, LLC, Dallas, Texas
  - UT Southwestern Medical Center, Dallas, Texas
  - North Texas Center for Clinical Research, Frisco, Texas
  - UTMB Department of Dermatology, Galveston, Texas
  - University of Texas Health Science Center at Houston, Houston, Texas
  - Arthritis & Osteoporosis Clinic, Waco, Texas
  - Velocity Clinical Research Waco, Waco, Texas
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - Open Door Clinical Research, Blacksburg, Virginia
  - West End Dermatology Associates, Richmond, Virginia
- Argentina (17):
  - CINME - Centro De Investigaciones Metabolicas, CABA, Buenos Aires
  - Centro de Investigaciones Medicas Mar del Plata, Mar del Plata, Buenos Aires
  - Instituto de Investigaciones Clinicas Quilmes, Quilmes, Buenos Aires
  - Centro de Investigaciones San Miguel, San Miguel, Buenos Aires
  - APRILLUS Asistencia e Investigacion, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Fundacion Respirar, Buenos Aires, Ciudad Autonoma Buenos Aires
  - Consultorio Alto Dorrego, Villa Nueva, Mendoza Province
  - Instituto CAICI, Rosario, Santa Fe Province
  - Clinica Mayo de Urgencias Medicas Cruz Blanca SRL, San Miguel de Tucumán, Tucumán Province
  - Centro de Investigaciones Medicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Investigaciones Clinicas Tucuman, San Miguel de Tucumán, Tucumán Province
  - Hospital Italiano de La Plata, Buenos Aires
  - Hospital Italiano de Buenos Aires, Ciudad Autonoma Buenos Aires
  - Centro Privado de Medicina Familiar - Mind Out Research, Ciudad Autonoma Buenos Aires
  - Clinica Adventista Belgrano, Ciudad Autonoma Buenos Aires
  - Instituto de Reumatologia, Mendoza
  - CER San Juan Centro Polivalente de Asistencia e Inv. Clinica, San Juan
- Belgium (2):
  - UZ Leuven, Leuven, Vlaams-Brabant
  - Universitair Ziekenhuis Gent, Ghent
- Brazil (18):
  - HUWC - UFC - Hospital Universitário Walter Cantídio - Universidade Federal do Ceará, Fortaleza, Ceará
  - CEDOES - Diagnóstico e Pesquisa, Vitória, Espírito Santo
  - Clínica SER da Bahia, Salvador, Estado de Bahia
  - L2IP - Instituto de Pesquisas Clínicas Ltda., Brasília, Federal District
  - IPC MT Instituto de Pesquisas Clinicas do Mato Grosso, Santo Ângelo, Mato Grosso
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - CMiP - Centro Mineiro de Pesquisa, Juiz de Fora, Minas Gerais
  - Instituto Brasil de Pesquisa Clínica-IBPCLIN S/A, Rio de Janeiro, Rio Do Janeiro
  - IDERJ - Instituto de Dermatologia e Estética do Brasil Ltda, Rio de Janeiro, Rio Do Janeiro
  - Hospital Bruno Born, Lajeado, Rio Grande do Sul
  - Hospital de Clínicas de Porto Alegre, Porto Alegre, Rio Grande do Sul
  - Nucleo de Pesquisa Clinica do Rio Grande do Sul, Porto Alegre, Rio Grande do Sul
  - LMK Serviços Médicos S/S Ltda, Porto Alegre, Rio Grande do Sul
  - Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul
  - CEMEC - Centro Multidisciplinar de Estudos Clínicos, São Bernardo do Campo, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica e Serviços Médicos, São Paulo, São Paulo
  - A2Z Clinical Centro Avancado de Pesquisa Clinica, Valinhos, São Paulo
  - RDSS Ricardo Diaz Scientific Solution, São Paulo
- Bulgaria (9):
  - DCC-1-Sevlievo EOOD, Sevlievo, Gabrovo
  - DCC 'Sveti Georgi' EOOD, Haskovo
  - Medical center Medconsult Pleven OOD, Pleven
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - DCC 1 - Ruse, EOOD, Rousse
  - Ambulatory for Specialized Medical Help - skin and venereal diseases, Sofia
  - DCC 'Alexandrovska', EOOD, Sofia
  - DCC Focus 5 - MEOH OOD, Sofia
  - Military Medical Academy - MHAT - Sofia, Sofia
- Canada (5):
  - Laser Rejuvenation Clinics, Inc., Calgary, Alberta
  - Laster Rejuvenation Clinics Edmonton D.T. Inc., Edmonton, Alberta
  - Medicor Research Inc, Greater Sudbury, Ontario
  - Dermatology Ottawa Research Centre, Ottawa, Ontario
  - DIEX Recherche Sherbrooke Inc., Sherbrooke, Quebec
- Chile (7):
  - Centro Medico SkinMed, Las Condes
  - Dermacross, Santiago
  - BioMedica Research Group, Santiago
  - CeCim Biocinetic, Santiago
  - CIEC - Centro Internacional de Estudios Clínicos, Santiago
  - Clinical Research Chile SpA., Valdivia
  - Oncocentro APYS, Viña del Mar
- China (26):
  - Beijing Tongren Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Affiliated Hospital of Fujian Medical University, Fuzhou, Fujian
  - Dongguan People's Hospital, Dongguan, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Second People's Hospital, Shenzhen, Guangdong
  - Zhongshan TCM Hospital, Zhongshan, Guangdong
  - Sun Yat-Sen Memorial Hospital, Sun Yat-Sen University, Guangzhou, Guangzhou
  - Nanyang First People's Hospital, Nanyang, Henan
  - Henan Provincial People's Hospital, Zhengzhou, Henan
  - Xiangya Hospital of Central South University, Changsha, Hu'nan
  - The second Xiangya Hospital of Central South University, Changsha, Hu'nan
  - The First Affiliated Hospital of Baotou Medical College, Baotou, Inner Mongolia
  - Hospital for Skin Diseases, Chinese Academy of Medical Sciences, Nanjing, Jiangsu
  - Affiliated Hospital of Jiangsu University, Zhenjiang, Jiangsu
  - The First Hospital of Jilin University, Changchun, Jilin
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Ruijin Hospital of Shanghai Jiaotong University School of Medicine, Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University, Shanghai, Shanghai Municipality
  - Shanghai Skin Disease Hospital, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Kunming Medical University, Kunming, Yunnan
  - The First Affiliated Hospital of Zhejiang University school of medicine, Hangzhou, Zhejiang
  - Hangzhou First People's Hospital, Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang
- Colombia (4):
  - Centro de Investigacion Medico Asistencial S.A.S, Barranquilla, Atlántico
  - Healthy Medical Center, Zipaquirá, Cundinamarca
  - Servimed S.A.S., Bucaramanga, Santander Department
  - Centro de Investigacion en Reumatologia y Especialidades Medicas SAS. CIREEM, Bogotá
- France (11):
  - CHU Nice - Hopital de l Archet, Nice, Alpes Maritimes
  - Hôpital de la Timone, Marseille, Bouches-du-Rhône
  - CHU de Caen - Hopital de la Cote de Nacre, Caen, Calvados
  - CHU Besançon - Hôpital Jean Minjoz, Besançon, Doubs
  - Hopital Larrey, Toulouse, Haute Garonne
  - Hôpital Privé d'Antony, Antony, Hauts De Seine
  - Hopital Saint Eloi, Montpellier, Herault
  - Hopital Claude Huriez - CHU Lille, Lille, Nord
  - Hôpital Saint-Louis, Cedex 10, Paris
  - Hopital Edouard Herriot - CHU Lyon, Lyon, Rhone
  - Hopital Tenon, Paris
- Germany (17):
  - Universitaetsklinikum Heidelberg, Heidelberg, Baden-Wurttemberg
  - Universitaetsklinikum Tuebingen, Tübingen, Baden-Wurttemberg
  - Universitaetsklinikum Erlangen, Erlangen, Bavaria
  - Klinikum rechts der Isar der TU Muenchen, Munich, Bavaria
  - Universitaetsklinikum Regensburg, Regensburg, Bavaria
  - Universitaetsklinikum Wuerzburg, Würzburg, Bavaria
  - Fachklinik Bad Bentheim Dermatologie, Bad Bentheim, Lower Saxony
  - Elbekliniken Buxtehude GmbH, Buxtehude, Lower Saxony
  - Klinikum Oldenburg AoeR, Oldenburg, Lower Saxony
  - Universitaetsklinikum Aachen AoeR, Aachen, North Rhine-Westphalia
  - Universitaetsklinikum Bonn AoeR, Bonn, North Rhine-Westphalia
  - Universitaetsklinikum Duesseldorf AoeR, Düsseldorf, North Rhine-Westphalia
  - Universitaetsklinikum Muenster, Münster, North Rhine-Westphalia
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden, Saxony
  - Universitaetsklinikum Halle (Saale), Halle, Saxony-Anhalt
  - Universitaetsklinikum Schleswig-Holstein - Campus Kiel, Kiel, Schleswig-Holstein
  - Charité - Campus Charité Mitte, Berlin
- Pecsi Tudomanyegyetem, Pécs, Hungary
- Italy (8):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi IRCCS, Bologna
  - Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Presidio Spedali Civili), Brescia
  - Università degli studi di Firenze, Florence
  - IRCCS Ospedale Policlinico San Martino, Genova
  - Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico, Milan
  - Ospedale San Raffaele, Milan
  - Azienda Ospedaliera Universitaria Policlinico 'Federico II', Napoli
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma
- Japan (30):
  - JCHO Chukyo Hospital, Nagoya, Aichi-ken
  - NHO Nagoya Medical Center, Nagoya, Aichi-ken
  - Fujita Health University Hospital, Toyoake-shi, Aichi-ken
  - Aomori Prefectural Central Hospital, Aomori, Aomori
  - Juntendo University Urayasu Hospital, Urayasu-shi, Chiba
  - University of Fukui Hospital, Yoshida-gun, Fukui
  - Hospital of the University of Occupational and Environmental Health, Kitakyushu-shi, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Kakogawa Central City Hospital, Kakogawa-shi, Hyōgo
  - Kita Harima Medical Center, Ono-shi, Hyōgo
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - St. Marianna University Hospital, Kawasaki-shi, Kanagawa
  - Yokohama City University Medical Center, Yokohama, Kanagawa
  - Yokohama City University Hospital, Yokohama, Kanagawa
  - NHO Yokohama Medical Center, Yokohama, Kanagawa
  - Kumamoto University Hospital, Kumamoto, Kumamoto
  - Tohoku University Hospital, Sendai, Miyagi
  - Nagasaki University Hospital, Nagasaki, Nagasaki
  - Niigata University Medical & Dental Hospital, Niigata, Niigata
  - Japanese Red Cross Okayama Hospital, Okayama, Okayama-ken
  - NHO Osaka Minami Medical Center, Kawachinagano-shi, Osaka
  - Daini Osaka Police Hospital, Osaka, Osaka
  - Kindai University Hospital, Osakasayama-shi, Osaka
  - Osaka University Hospital, Suita-shi, Osaka
  - Takatsuki Red Cross Hospital, Takatsuki-shi, Osaka
  - Shiga University of Medical Science Hospital, Ōtsu, Shiga
  - Shimane University Hospital, Izumo-shi, Shimane
  - Teikyo University Hospital, Itabashi-ku, Tokyo-To
  - Showa University East Hospital, Shinagawa-ku, Tokyo-To
  - Wakayama Medical University Hospital, Wakayama, Wakayama
- Mexico (7):
  - Centro de investigacion medica y reumatologia, Guadalajara, Jalisco
  - Centro de Investigacion Clínica GRAMEL S.C, Mexico City, Mexico City
  - Clinstile, S.A. de C.V., Mexico City, Mexico City
  - Consultorio Privado Dr. Miguel Cortes Hernandez, Cuernavaca, Morelos
  - Medical Care & Research SA de CV, Mérida, Yucatán
  - Derma Norte del Bajio S.C., Aguascalientes
  - Investigacion y Biomedicina de Chihuahua, S.C., Chihuahua City
- Peru (2):
  - ACQ MEDIC SAC - Centro de Investigacion Clinica Inmunoreumatologia, Lima
  - Invest Clinicas Sac Inst de Ginecologia y Reproduccion, Lima
- Philippines (9):
  - The Medical City Clark, Mabalacat, Pampanga
  - Cebu Doctors University Hospital, Cebu City
  - Mary Mediatrix Medical Center, Lipa City
  - Medical Center Manila, Manila
  - Philippine General Hospital, Manila
  - Jose R. Reyes Memorial Medical Center, Manila
  - St. Luke's Medical Center, Quezon City
  - Far Eastern University - Dr. Nicanor Reyes Medical Foundation, Quezon City, Metro Manila
  - Ilocos Training and Regional Medical Center, San Fenando, La Union
- Poland (11):
  - DERMEDIC Jacek Zdybski, Kielce
  - SPZOZ Szpital Uniwersytecki w Krakowie, Krakow
  - Promed P.Lach R.Glowacki spolka jawna, Centrum Medyczne PROMED, Krakow
  - Specjalistyczny Gabinet Dermatologiczny Aplikacyjno-Badawczy Marek Brzewski, Krakow
  - MT Medic Specjalistyczna Praktyka Lekarska Tomasz Stapinski, Krosno
  - Dermoklinika Centrum Medyczne SC M Kierstan J Narbutt A Lesiak, Lodz
  - Kliniczny Szpital Wojewodzki nr 1 im.F.Chopina, Rzeszów
  - MICS Centrum Medyczne Warszawa, Warsaw
  - Szpital Kliniczny Dzieciatka Jezus, Warsaw
  - Royalderm, Warsaw
  - Cityclinic Przychodnia Lekarsko-Psychologiczna Matusiak Spółka Partnerska, Wroclaw
- Portugal (5):
  - Centro Hospitalar e Universitário de Coimbra, E.P.E (HUC), Coimbra
  - Hospital de Egas Moniz, Lisbon
  - Hospital CUF Descobertas, Lisbon
  - Centro Hospitalar Universitártio do Porto, E.P.E., Porto
  - Unidade Local de Saúde do Alto Minho, E.P.E., Viana do Castelo
- Puerto Rico (2):
  - Dr. Samuel Sanchez PSC, Caguas
  - GCM Medical Group PSC - Hato Rey, San Juan
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Center, Riyadh
  - King Saud University, Riyadh
- Serbia (4):
  - Institute of Rheumatology, Belgrade
  - University Clinical Center of Serbia, Belgrade
  - University Clinical Center Kragujevac, Kragujevac
  - Clinical Center of Vojvodina, Novi Sad
- Slovakia (2):
  - Artromac n.o., Košice
  - Narodny ustav reumatickych chorob, Piešťany
- South Korea (6):
  - Korea University Ansan Hospital, Ansan-si, Gyeonggi-do
  - Ajou University Hospital, Suwon, Gyeonggi-do
  - Chonnam National University Hospital, Gwangju
  - Severance Hospital, Yonsei University Health System, Seoul
  - Hanyang University Seoul Hospital, Seoul
  - The Catholic University of Korea, Seoul St. Mary's Hospital, Seoul
- Spain (10):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario Rio Hortega, Valladolid, Cantabria
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Universitario Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitari Vall d'Hebron - VHIR, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Reina Sofia, Córdoba
  - Hospital Universitario Virgen del Rocio, Seville
- Karolinska Universitetssjukhuset - Solna, Stockholm, Sweden
- Switzerland (3):
  - Universitaetsspital Zuerich, Zurich-Flughafen, Canton of Zurich
  - Centre Hospitalier Universitaire Vaudois (CHUV), Lausanne
  - Kantonsspital St. Gallen, Sankt Gallen
- Taiwan (5):
  - Changhua Christian Medical Foundation Changhua Christian Hospital, Changhua
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (4):
  - Whipps Cross University Hospital, London, Greater London
  - Manchester Royal Infirmary, Manchester, Greater Manchester
  - Queen Elizabeth Hospital, Birmingham, West Midlands
  - Chapel Allerton Hospital, Leeds, West Yorkshire

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org